CLINICAL TRIAL: NCT01182064
Title: Relationship of Echocardiographic and Coronary Angiographic Findings in Patients With Acute Myocardial Infarction Secondary to Penetrating Cardiac Trauma
Brief Title: Acute Myocardial Infarction by Penetrating Cardiac Trauma
Status: Completed | Type: Observational
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Wilfredy Castano, Antioquia University Student
Other Study IDs: WCJWJ1
Record Dates: First submitted 2010-08-13; First posted 2010-08-16 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2007-03

CONDITIONS: Myocardial Infarction
Keywords: Heart injuries; Posttraumatic myocardial infarction; Echocardiography; Coronary angiography
MeSH Terms: conditions — Myocardial Infarction; Heart Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non infarct
- Posttraumatic acute myocardial infarct without coronary injury
- Posttraumatic acute myocardial infarct with coronary injury

SUMMARY:
Patients with a cardiac stab wound could be complicated by a posttraumatic acute myocardial infarction (PAMI). Traditionally, the investigators can explain it by the occlusion of a coronary artery; but the PAMI isn´t constantly related with coronary artery injuries or their damage in the cardiac injury repair. The investigators objectives are to know the PAMI incidence, make an approximation to PAMI pathophysiology, and propose management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Heart stab Injury

Exclusion Criteria:

* Previous cardiac injuries, coronary artery disease with previous diagnostic, previous coronary angiography (for any indication)

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included patients admitted to the emergency department of the San Vicente de Paul University Hospital with a penetrating stab cardiac injury without previous injuries
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2007-04; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Posttraumatic acute myocardial infarct | 2 days

SECONDARY OUTCOMES:
Posttraumatic acute myocardial infarct without coronary injury | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos H Morales, MD, MSc, Study Director — Antioquia University
Locations (1):
- San Vicente de Paul Hospital, Medellín, Antioquia, Colombia

REFERENCES:
- [Derived] Castano W, Morales CH, Senior JM, Benjumea WY, Sanchez J. Relationship of echocardiographic and coronary angiographic findings in patients with acute myocardial infarction secondary to penetrating cardiac trauma. J Trauma Acute Care Surg. 2012 Jul;73(1):111-6. doi: 10.1097/TA.0b013e318256a0d8. PMID 22743380